CLINICAL TRIAL: NCT06488105
Title: Initiating Preventive Care for Hyperlipidemia in the Emergency Department: The EMERALD (Emergency Medicine Cardiovascular Risk Assessment for Lipid Disorders) Trial
Brief Title: Emergency Medicine Cardiovascular Risk Assessment for Lipid Disorders Trial
Acronym: EMERALD RCT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00104057; 1K23HL169929-01A1 (NIH)
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-03

CONDITIONS: Lipid Disorder; Hypercholesterolemia; Cardiovascular Diseases; Atherosclerosis
Keywords: hyperlipidemia; cardiovascular disease; atherosclerotic cardiovascular disease
MeSH Terms: conditions — Lipid Metabolism Disorders; Hypercholesterolemia; Cardiovascular Diseases; Atherosclerosis; Hyperlipidemias | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: 130 Emergency Department patients will be randomized with chest pain 1:1 to Emergency Medicine Cardiovascular Risk Assessment for Lipid Disorders (EMERALD) or usual care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Emergency Medicine Cardiovascular Risk Assessment for Lipid Disorders (EMERALD) arm (Experimental): In the EMERALD arm, care will vary by risk level: (1) patients with known atherosclerotic cardiovascular disease (ASCVD) will qualify for a high-intensity statin (rosuvastatin 40 mg daily) and referral to cardiology for secondary prevention, (2) patients with low-density lipoprotein cholesterol (LDL-C) ≥190 mg/dL will receive a high-intensity statin and a cardiology referral for primary prevention, and (3) for the remaining patients, Emergency Department providers will calculate 10-year ASCVD risk using the Pooled Cohort Equations. These patients will be categorized as (3A) high risk patients (10-year risk ≥20%) who will receive a high-intensity statin and a cardiology referral and (3B) moderate risk patients (10-year risk ≥7.5% but <20% or those with known diabetes and 10-year risk <20%) who will receive a moderate-intensity statin (rosuvastatin 10 mg daily) and a primary care referral. EMERALD patients will also receive healthy lifestyle counseling.
  Interventions: Drug: Statin (rosuvastatin 10 or 40 mg daily, depending on risk); Behavioral: Healthy Lifestyle Counseling; Other: Outpatient Followup
- Usual Care Arm (Active Comparator): Patients in the usual care arm will receive the current standard of care, which consists of primary care referral and no Emergency Department statin prescription. They will also receive healthy lifestyle counseling.
  Interventions: Behavioral: Healthy Lifestyle Counseling; Other: Outpatient Followup

INTERVENTIONS:
Drug: Statin (rosuvastatin 10 or 40 mg daily, depending on risk) — moderate- or high-intensity statin (either rosuvastatin 10 mg daily or rosuvastatin 40 mg daily)
  Other Names: Crestor
  Arms: Emergency Medicine Cardiovascular Risk Assessment for Lipid Disorders (EMERALD) arm
Behavioral: Healthy Lifestyle Counseling — Healthy lifestyle counseling based off the American Heart Association's Life Essential 8 framework
Other: Outpatient Followup — Emergency Medicine Cardiovascular Risk Assessment for Lipid Disorders (EMERALD) intervention patients will receive either cardiology or primary care referral (depending on risk level) and usual care patients will receive a primary care referral

SUMMARY:
Emergency Medicine Cardiovascular Risk Assessment for Lipid Disorders (EMERALD) is a protocolized intervention based on American College of Cardiology/American Heart Association and US Preventive Services Task Force guidelines designed to initiate preventive cardiovascular care for emergency department patients being evaluated for acute coronary syndrome. The overarching goals of this proposal are to (1) determine the efficacy of EMERALD at lowering low-density lipoprotein cholesterol (LDL-C) and non high-density lipoprotein cholesterol (non-HDL-C) among at-risk Emergency Department (ED) patients who are not already receiving guideline-directed outpatient preventive care and (2) inform our understanding of patient adherence and determinants of implementation for ED-based cardiovascular disease prevention strategies.

DETAILED DESCRIPTION:
EMERALD involves (1) ordering an ED lipid panel, (2) calculating 10-year atherosclerotic cardiovascular disease (ASCVD) risk, (3) prescribing a moderate- or high-intensity statin, (4) providing healthy lifestyle counseling, and (5) bridging patients to ongoing outpatient preventive care (primary care or cardiology, depending on risk level).

We hypothesize that EMERALD will be associated with lower LDL-C and non-HDL-C at 30- and 180-days vs. usual care. The primary outcome will be percent change in LDL-C at 30-days. Secondary outcomes include percent change in LDL-C at 180-days and non-HDL-C at 30- and 180-days. We will randomize 130 ED patients with possible acute coronary syndrome 1:1 to EMERALD or usual care, which will provide 90% power with a two-sided alpha of 0.05 to demonstrate a 10% difference in percent change in LDL-C at 30-days between arms.

ELIGIBILITY:
Inclusion Criteria

1. Evaluation for Acute Coronary Syndrome
2. Age 40-75 Years
3. 10-year Atherosclerotic Cardiovascular Disease (ASCVD) Risk ≥7.5% or Known Diabetes or

Known ASCVD:

1. Myocardial Infarction
2. Unstable Angina
3. Percutaneous Coronary Intervention
4. Coronary Artery Bypass Graft
5. Stroke
6. Transient Ischemic Attack
7. Peripheral Artery Disease

Exclusion Criteria

1. ST-Segment Elevation Myocardial Infarction (STEMI) Activation
2. ST Depression >1 mm in Contiguous Leads
3. On a Lipid Lowering Agent (Statin, PCSK9 Inhibitor, Bempedoic Acid, Ezetimibe, Inclisiran, etc.)
4. Inability to Return for 30-day Follow-up
5. Unstable Vitals (Systolic blood pressure <90, HR >120 or <50, oxygen saturation <90%)
6. Statin Intolerance
7. Any Resulted High-Sensitivity Troponin I ≥100 ng/L
8. End-stage renal disease (ESRD) and/or glomerular filtration rate (GFR) <30 mL/min/1.73 m2
9. Liver Cirrhosis
10. Pregnancy
11. Anticipated Hospitalization
12. Life Expectancy <1 Year
13. Transfer from Another Hospital
14. Prisoner
15. Non-English Speaking

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Percent change in low-density lipoprotein cholesterol (LDL-C) at 30 days | Index ED encounter through 30 days (-3, +11 days)
  Percent change in LDL-C from the index Emergency Department (ED) encounter through 30 days

SECONDARY OUTCOMES:
Percent change in LDL-C at 180 days. | Index ED encounter through 180 days (+/- 15 days)
  Percent change in LDL-C from the index ED encounter through 180 days
Percent change in non high-density lipoprotein cholesterol (non-HDL-C) at 30 days | Index ED encounter through 30 days (-3, +11 days)
  Percent change in non-HDL-C from the index ED encounter through 30 days
Percent change in non-HDL-C at 180 days | Index ED encounter through 180 days (+/- 15 days)
  Percent change in non-HDL-C from the index ED encounter through 180 days
Proportion of patients with outpatient clinic follow-up at 30 days | Index ED encounter through 30 days (-3, +8 days)
  Did the patient follow-up with the recommended outpatient care team?
Proportion of patients with statin prescription pick-up | Index ED encounter through 10 days
  Did the patient pick-up their statin prescription from the pharmacy?
Qualitative barriers and facilators | 30 days (+30 days) after the index ED encounter
  Qualitative interviews to determine facilitators and barriers to the Emergency Medicine Cardiovascular Risk Assessment for Lipid Disorders (EMERALD) program

CONTACTS AND LOCATIONS:
Overall Officials: Nick Ashburn, Principal Investigator — n.ashburn@wakehealth.edu
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No